CLINICAL TRIAL: NCT02357524
Title: A Single Center, Open-label Study to Evaluate the Effects of a Single 1200mg IV Dose of Oritavancin on the Results of Multiple Coagulation Tests in Healthy Volunteers
Brief Title: Oritavancin on the Results of Multiple Coagulation Tests in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Collaborators: Christchurch Clinical Studies Trust Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MDCO-ORI-14-01
Record Dates: First submitted 2015-01-27; First posted 2015-02-06 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers
Keywords: Effects on coagulation tests in healthy volunteers
MeSH Terms: interventions — oritavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oritavancin (Experimental): Subject will receive a single oritavancin dose of 1200 mg in 1000 mL of D5W administered as a constant rate IV infusion over 3 hours via a single dedicated peripheral venous line.
  Interventions: Drug: Oritavancin

INTERVENTIONS:
Drug: Oritavancin

SUMMARY:
The study will determine the magnitude and duration (time to resolution i.e., returning to normal ranges) of elevations in the following coagulation test results after a single 1200 mg dose of oritavancin: Prothrombin Time/International Normalized Ratio (PT/INR), Activated clotting time (ACT), Activated Partial Thromboplastin Time (APTT), Chromogenic Factor Xa Assay, D-dimer, Silica Clot Time and Dilute Russell's Viper Venom Time (DRVVT).

DETAILED DESCRIPTION:
Oritavancin has been approved in the United States for the treatment of adult patients with acute bacterial skin and skin structure infections (ABSSSIs) caused or suspected to be caused by susceptible isolates of designated Gram-positive microorganisms.

Antibiotics of this class (lipoglycopeptide and lipopeptide antibiotics) artificially prolong phospholipid-dependent coagulation tests such as prothrombin time (PT) and activated partial thromboplastin time (aPTT) by binding to and preventing the action of the phospholipid reagents needed to activate coagulation.

Because precipitation of oritavancin has been shown to occur in human plasma at concentrations as low as 50 μg/mL in vitro, a relevant approach to further elucidate the full range of effects of oritavancin plasma concentrations on coagulation testing would be to conduct a clinical study in healthy volunteers in which coagulation tests are monitored following a single 3 hour infusion of 1200 mg oritavancin. The data from this study will help inform physicians about how to manage patients who require coagulation monitoring in the setting of treatment with oritavancin.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to provide written informed consent before initiation of any study-related procedures.
2. Subject is a healthy male or female adult between 18 and 65 years of age, inclusive.
3. Subject has a body mass index (BMI) < 45 kg/m2.
4. Subject is in good health based on medical history and physical examination findings and has no clinically meaningful safety laboratory abnormalities (CBC, blood chemistry, and urinalysis) or 12-lead ECG results, as assessed by the Principal Investigator (PI).
5. Vital signs (BP, pulse and temperature) measured at screening/baseline must be within the following ranges: SBP ≥90 to ≤150 mm Hg, DBP ≥45 to ≤90 mm Hg; Heart Rate ≥ 45 to ≤90 bpm (taken after resting in a supine position for at least 5 minutes).
6. Female subject is surgically sterile, postmenopausal, or, if of childbearing potential, agrees to use at least 2 acceptable methods of birth control (e.g. prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, barrier methods, abstinence) or male partner sterilization alone for the duration of the study until 60 days after study drug administration.

Exclusion Criteria:

1. Has any condition, including findings in the medical history or in prestudy assessments that constitutes a risk or a contraindication for the participation in the study or completing the study.
2. Any coagulation test results that are outside of the normal range at Screening.
3. Any of the following coagulation tests results that are outside of the normal range at Baseline (Pre-Dose): Prothrombin Time/International Normalized Ratio (PT/INR), Activated clotting time (ACT), Activated Partial Thromboplastin Time (APTT).
4. Positive breath test for alcohol and/or positive urine test for drugs of abuse at Screening.
5. Has a history or presence of alcohol/drug abuse within 2 years. Alcohol abuse is defined as regularly consuming >3 units/day (21 units per week for men), >2 units/day (14 units/week) for women. A unit is defined as a can of 4% beer (330 mL), approximately 190 mL of 6-7% beer (malt liquor), a glass of 40% spirits (30 mL), a glass of wine (100 mL).
6. Blood or plasma donation within past 2 months.
7. History of hypersensitivity to drugs with a similar chemical structure (i.e. glycopeptide antibiotics) to the investigational product or any of its excipients.
8. Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 90 days prior to enrollment and/or unwilling to allow at least two months before participation in another drug trial following the current trial.
9. Treatment with any prescription or OTC drugs, within 2 weeks or five half-lives, whichever is longer, or herbal nutritional supplements within 2 weeks of screening, with the exception of acetaminophen/paracetamol for minor headache. Subjects will not be allowed to receive medications for the duration of the study (except the abovementioned acetaminophen/paracetamol). Birth control or other hormone replacement is also permitted as long as it has been taken at a stable dose for at least three months before the Screening Visit and remains stable for the duration of the study.
10. Females who are pregnant or nursing or who have a positive pregnancy test result at screening.
11. Males who are unwilling to practice abstinence or use an acceptable method of birth control during the entire study period (i.e. condom with spermicide, where locally available).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Time to resolution of elevations in coagulation test results | up to 120 hours
  Time to resolution of elevations in PT/INR, ACT, APTT, Chromogenic Factor Xa level, D-dimer, Silica Clot Time and DRVVT value will be descriptively summarized for each assay. If appropriate, two-sided 95% confidence interval for the median time will also be provided.

SECONDARY OUTCOMES:
Changes from baseline in coagulation test results | up to 120 hours
  Changes from baseline in PT/INR, ACT, APTT, Chromogenic Factor Xa level, D-dimer, Silica Clot Time and DRVVT value will be summarized for each assay at each post-baseline time point. Two-sided 95% confidence interval for the changes will also be provided. The number and percentage of subjects having coagulation test values outside normal ranges will also be summarized for each assay at each post-baseline time point.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Melinta Therapeutics, Inc.
Locations (1):
- Christchurch, New Zealand